CLINICAL TRIAL: NCT05399407
Title: Randomized Controlled Trial PRALIMAP-CINeCO: Comparison of Health E-coaching Versus Referral to the Usual Care System for Overweight and Obese Young Adults
Brief Title: PRALIMAP-CINeCO: Comparison of Health E-coaching Versus Referral to the Usual Care System
Acronym: PRALIMAPCINeCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other); Cnam-ISTNA (Unknown)
Responsible Party: Principal Investigator, Yacoubou OMOROU, Principal Investigator, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021PI178
Record Dates: First submitted 2022-05-03; First posted 2022-06-01 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Overweight and Obesity
Keywords: E-coaching; Usual Care System; young adults
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Experimental group: health e-coaching Control group: standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: health e-coaching (Experimental): * Personalised and secure access to the health e-coaching platform for 12 months.
  * Follow-up by professionals who are specialized in the subject matter (at a distance): a psychologist, a dietician and a teacher of adapted physical activity.
  * Personalised activities offered to each young adult throughout their follow-up: synchronous and asynchronous activities (video, animation, quizzes, etc.), individual and collective on different themes (expression of emotions, my weight and me, eating well to start with, my image and me, making choices, my way of moving, etc.). The personalisation of the activities will be done in consultation between the professionals and the young adult according to the needs expressed and identified.
  Interventions: Other: Health e-coaching
- Control group: Usual Care System (No Intervention): Control group : - Referral to health professionals in the health care system and, in priority, to the GP declared by the young adult.
  - Transmission of the data collected during follow-up visit No. 3 / 0 (T3/T0) to the GP with relay for the implementation of a care plan.

INTERVENTIONS:
Other: Health e-coaching — Management of overweight / obesity
  Arms: Experimental group: health e-coaching

SUMMARY:
This study involves young adults from the PRALIMAP-INES trial and student volunteers from the University of Lorraine, who are overweight or obese.

For young adults from the PRALIMAP-INES trial, the proposed research is a continuation of the PRALIMAP-CINeCO research (part 1).

For students at the University of Lorraine, the proposed research is aimed at volunteer students who are overweight or obese, via the University of Lorraine's Student Health Service (SSE).

Young adults and overweight or obese students not receiving medical care at the time of the inclusion visit (4th measurement time for PRALIMAP-INES participants and 1st time for others) will be offered the chance to take part in a randomized trial comparing the acceptability of health e-coaching versus referral to standard care.

Experimental group: health e-coaching Control group: usual care system

Primary objective : To determine the effectiveness of an e-health coaching intervention using new technologies that promotes changes in eating and physical activity behavior in overweight and obese young adults aged 20, an intervention targeting the development of autonomous self-regulation.

Secondary objectives :

1. Determine the acceptability of health e-coaching: acceptability of new technologies (container), acceptability of personalized health e-coaching (content).
2. Determine the effectiveness of health e-coaching on the criteria of corpulence (BMI; body composition), changes in eating behaviors (TCA), emotion management skills and social interaction skills.
3. Evaluate the benefit of health e-coaching alone or combined with the previous intervention received in the PRALIMAP-INÈS trial on primary and secondary endpoints.
4. Evaluate and compare participation in a health promotion program over two life periods (adolescence and young adulthood) for young adults from the PRALIMAP-INÈS trial.
5. Evaluate the effectiveness of health e-coaching (reinforcement of autonomous self-regulation and changes in eating behaviors and physical activity practices/time spent sitting) according to the dose of intervention received by young adults (received-treatment analysis).
6. Determine the cost-efficiency and cost-utility ratios by means of a medico-economic evaluation based on the incremental cost of the e-coaching intervention in relation to the usual care offered by the health care system (ICER: Incremental Cost-Effectiveness Ratio).

ELIGIBILITY:
Inclusion Criteria:

Among the young adults who agreed to participate in follow-up visit (T3) in the PRALIMAP-CINeCO trial (Part 1), the inclusion criteria for the inclusion criteria for the proposed research are as follows:

* Person having received complete information on the organization of the research and not and who did not object to their participation and to the use of their data to participate and to use their data
* Have agreed to complete the pre-test questionnaire prior to/at the follow-up visit (T3)
* Have agreed to the anthropometric measurements without invasive intervention performed at the follow-up visit (Q3)
* Have a BMI greater than 25kg/m² (Cole et al. 2000) or a percentage of body fat mass greater than or equal to 20% for men and greater than or equal to 33% for women, depending on age and greater than or equal to 33% for women and not receiving medical medical care for this situation
* Agree to participate in the follow-up
* Accepting the health e-coaching/orientation to routine care
* Affiliated to a social security system or beneficiary of such a system
* Reside in France

Among the students who agreed to participate, through the Student Health Service of the University of Lorraine, the inclusion criteria for the proposed research are as follows:

* Person having received complete information on the organization of the research and not and who did not object to their participation and to the use of their data to participate and to use their data
* Have agreed to complete the pre-test questionnaire prior to/at the follow-up visit (T0)
* Have agreed to the anthropometric measurements without invasive intervention performed at the follow-up visit (T0)
* Have a BMI greater than 25kg/m² (Cole et al. 2000) or a percentage of body fat mass greater than or equal to 20% for men and greater than or equal to 33% for women, depending on age and greater than or equal to 33% for women and not receiving medical medical care for this situation
* Agree to participate in the follow-up
* Accepting the health e-coaching/orientation to routine care
* Affiliated to a social security system or beneficiary of such a system
* Reside in France
* Be of legal age (18 years or older)
* Be a student at the Université de Lorraine

Exclusion Criteria:

If the follow-up visit n°3 (T3) during the PRALIMAP-CINeCO trial (1st part) or the inclusion visit (T0 for University of Lorraine students), was completed, the non-inclusion criteria for the referral of young adults young adults (health e-coaching/current care) are as follows:

* Do not feel the need for coaching
* Be already being treated for overweight by a health professional specializing in the treatment of specialized in the treatment of overweight and obesity or a specialized specialized medical structure/service
* Do not agree to participate in the continuation of PRALIMAP-CINeCO
* Major person under a legal protection measure (guardianship, curatorship, safeguard of justice)
* Persons deprived of liberty by a judicial or administrative decision administrative decision Persons under psychiatric care in accordance with Articles L. 3212-1 and L. 3213-1 of the Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-01-09 (Estimated); Study Completion 2025-01-09 (Estimated)

PRIMARY OUTCOMES:
Evolution of the corpulence determined from the body mass index [BMI] | Before and after intervention, an average of 1 year
  Body Mass Index (BMI) indicates the ratio between your weight and your height in meters squared (kg/m^2)
Change of the eating behaviors | Before and after intervention, an average of 1 year
  Diet, tobacco and alcohol consumption (food frequency questionnaire)
Change of the physical activity practices | Before and after intervention, an average of 1 year
  Physical activity and sedentary behaviour (GPAQ)
Change of the Self-regulatory skills | Before and after intervention, an average of 1 year
  Adaptation strategy (BriefCOPE)
Change of the Self Efficacy Diet | Before and after intervention, an average of 1 year
  TESQ-E (Self-Efficacy Diet Questionnaire)

SECONDARY OUTCOMES:
Level of satisfaction | Study completion, an average of 1 year
  Satisfaction questionnaire
Change of the level of quality of Life | Before and after intervention, an average of 1 year
  Questionnaire EQ-5D-5L
Change of the Knowledge on nutrition and physical activity | Before and after intervention, an average of 1 year
  Questionnaire of knowledge on nutrition and physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No